CLINICAL TRIAL: NCT06714331
Title: The Effect of Acute Caffeine and Sodium Bicarbonate Supplementation on Upper and Lower Submaximal Resistance Training Performance
Brief Title: Caffeine and Sodium Bicarbonate Supplementation Effects on Resistance Training Performance
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, David George Behm, Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20241611
Record Dates: First submitted 2024-08-01; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Nutritional Supplementation; Resistance Training
Keywords: caffeine; sodium bicarbonate; strength; fatigue; resistance training
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, cross-over study design with 1 intervention (supplements) with 3 arms (caffeine, sodium bicarbonate, control placebo).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Separate investigator mixes the caffeine or sodium bicarbonate mixture solution. Other investigators conducting the data collection are blinded to the supplement or control mixture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Caffeine (Experimental): Caffeine supplement is consumed at 3 time points (120, 90 and 45 minutes prior to testing) with participants drinking 300mL of a caffeine and water solution at each time for a total consumed volume of 900mL .
  Caffeine concentration - 3mg/kg or 0.003g/kg
  Each solution has MiO Liquid Water Enhancer to mask the taste.
  Interventions: Dietary Supplement: Supplements
- Sodium bicarbonate (Experimental): Sodium bicarbonate supplement is consumed at 3 time points (120, 90 and 45 minutes prior to testing) with participants drinking 300mL of sodium bicarbonate solution at each time for a total consumed volume of 900mL.
  Sodium bicarbonate concentration - 0.3g/kg (Arm and Hammer brand)
  Each solution has MiO Liquid Water Enhancer to mask the taste.
  Interventions: Dietary Supplement: Supplements
- Control (Sham Comparator): Control solution is MiO + 300mL water at 3 time points (120, 90 and 45 minutes prior to testing) with participants drinking 300mL of control solution at each time for a total consumed volume of 900mL.
  Interventions: Dietary Supplement: Supplements

INTERVENTIONS:
Dietary Supplement: Supplements — Supplements provided to subjects 2 hours prior to testing and drank at 2 hours, 90 minutes and 45 minutes before testing.

SUMMARY:
This research aims to explore the effects of two supplements, caffeine and sodium bicarbonate, on acute (short-term) resistance training performance. The present study aims to assess the effects of caffeine and sodium bicarbonate supplementation on the number of repetitions, muscle activation, speed of movement, and fatigue during resistance training.

DETAILED DESCRIPTION:
The study will employ a randomized, double-blind, placebo-controlled, cross-over study design that examines the effect of caffeine and sodium bicarbonate on knee extension and bench press performance. Parameters include peak isoinertial force (1 repetition maximum: 1RM), rate of force development, movement velocity, number of repetitions to failure with a 10 repetition maximum (10RM) load, and electromyography (EMG) activity. The participants will complete three separate visits to the laboratory (1. placebo, 2. caffeine, and 3. sodium bicarbonate ingestion). With respect to the first visit, participants will sign a consent form and complete a health history questionnaire. Their respective anthropometric measurements will be taken, including height, weight, body mass index (BMI). Participants will then be introduced to the rate of perceived exertion scale for use during the trials. Blood lactate (Lactate Pro, Arkray, Kyoto, Japan) levels will be collected and analyzed from the index finger of the tested arm. Researchers will establish the 1RM for the bench press (upper-body) and knee extension (lower-body) exercises. The participants will complete a warm-up set of 8-10 repetitions at 50% of their body mass, followed by a 60-second rest period. The participants will then complete a second warm-up set of 3-5 repetitions with a 5-10 kg increase from the initial set, followed by another 60-second rest interval. the participants will then complete 2-3 repetitions with an additional 5-10 kg increase, followed by a rest for an additional 120 seconds. Each subsequent one-repetition attempt increased an additional 5-10 kg, followed by a 120-second rest period. The final attempt will be determined by repeating the steps illustrated above until the participants can no longer complete a single unassisted repetition with additional weight. This value will then be illustrated as the participant's 1RM and will be utilized to calculate exercise intensity for the two subsequent supplementation trials.

All testing will be performed within the laboratory. Participants are instructed to meet the following conditions 24-h before each experimental trial: (i) to avoid vigorous exercise, (ii) to adopt a similar diet and drink intake, (iii) to refrain from the consumption of alcohol, caffeine, and other stimulants.

Measures

For the knee extension measures, EMG activity will be collected from the mid-belly (midway between the anterior superior iliac spine to the superior edge of the patella) of the vastus lateralis and biceps femoris (midway between the gluteal fold and the popliteal space) of the non-dominant leg. Before participants perform the bench press, surface EMG recording electrodes will be placed approximately 3 cm apart over the proximal, lateral segment of the biceps brachii and over the lateral head of the triceps brachii. The distance of the biceps brachii electrodes from the acromion process and the distance of the triceps electrodes from the biceps electrodes will be recorded to ensure accurate replacement for subsequent tests. A thorough skin preparation for all electrodes will include shaving and removal of dead epithelial cells with abrasive pad around the designated areas, followed by cleansing with an isopropyl alcohol swab. EMG will be collected using a Biopac (Biopac Systems Inc.) data acquisition system at a sample rate of 2,000 Hz [impedance = 2 MΩ, common mode rejection ratio >110 dB min (50/60 Hz), noise >5 μV]. A bandpass filter (10-500 Hz) will be applied prior to digital conversion.

The root mean square (RMS) EMG will be monitored throughout the range of movements for both the bench press and knee extension. The mean RMS EMG will be normalized to the highest pre-test value and reported as a percentage.

A linear position transducer (Chronojump; Boscosystem, Barcelona, Spain) will be attached to the barbell to measure the excursion of the movement, time, and velocity. This device has been previously validated for velocity and power measurements.

Blood lactate levels will be measured with StatStrip Xpress Lactate (SSX) (Nova Biomedical, Waltham, Massachusetts, USA) prior to, during, and after the bench press and knee extension exercises to determine blood-lactate levels of the participants.

The participant's heart rate and rating of perceived exertion will be collected immediately after the completion of each set.

Intervention

During the subsequent three visits, participants will consume the placebo (dextrose), caffeine or sodium bicarbonate. A one week washout period will be allocated between visits. The same quantity will be used during both testing trials to ensure that the supplement is the only variable. The participants will spend 1 hour in a seated resting position after consuming the placebo or supplement. Participants will then utilize the same warm-up as the first visit, 8-10 repetitions at 50% of their body mass.

Testing Procedure

Using a 10RM load, participants will be instructed to complete as many repetitions as possible for each set (6 sets for each exercise) until they can no longer complete a repetition without assistance. Researchers will then record the number of repetitions participants complete during each set. The participant will then undergo a 60-second rest period between each set. After the participant completes the first exercise (e.g., six bench press or knee extension sets), they will undergo a 120-second rest period before beginning the same procedure on the next exercise (i.e., bench press or isoinertial knee extension resistance device). The order of bench press and knee extension exercises will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy, physically active males and females between 18-40 years of age with regular (minimum three times a week) resistance training experience for the last 6 months and regular caffeine intake (at least once a day).

Exclusion Criteria:

* recent musculoskeletal or musculotendinous injuries

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Bench press repetitions to failure | 45 minutes after last consumption of supplement or control drink solution.Order of bench press vs. knee extension is randomized.
  During familiarization participants 12 repetition maximum was calculated. After drinking supplement or control participants perform 6 sets of 12 repetition bench press maximum repetitions to failure.
  Outcome measure is the number of repetitions completed in each set of the 6 sets.
Knee extensions repetitions to failure | 45 minutes after last consumption of supplement or control drink solution. Order of bench press vs. knee extension is randomized.
  During familiarization participants 12 repetition maximum was calculated. After drinking supplement or control participants perform 6 sets of 12 knee extension maximum repetitions to failure.
  Outcome measure is the number of repetitions completed in each of the 6 sets.

SECONDARY OUTCOMES:
Blood lactate | Pre- (1 minute prior to ingestion of supplement solution) and post-tests (1 minute after each bout of bench press and knee extensions to failure). Each measure should take 5 seconds.
  Blood lactate obtained from index finger. Outcome measure is the millimoles of blood lactate at each testing time.
Heart rate | Heart rate (instantaneous feedback by monitor) will be recorded 10 seconds after every bench press and knee extension set in each condition/session (caffeine, sodium bicarbonate and control sessions).
  Heart rate detected by heart rate monitor instantaneously Outcome measure is the heart rate reported in beats per minute at each testing time.
Rating of perceived exertion | Recorded 20 seconds (response time = 2 seconds) after every bench press and knee extension set in each condition/session (caffeine, sodium bicarbonate and control sessions).
  Adapted Borg scale with scale from 1-10. Reporting should take 2 seconds upon each request by the investigator.
  Outcome measure is the participant's reported scale number at each testing time.
Electromyography (EMG) root mean square (Mean amplitude) | During every repetition to failure sets. Each set will take a maximum of 30 seconds. With fatigue from the repetitive 6 sets, the exercise and monitoring time will decrease.
  Surface EMG electrodes will be used to monitor muscle activation with every set of resistance training. The mean amplitude of the root mean square (RMS) of the EMG will be measured over the duration of each repetition. Filtering (band pass 5-500 Hz) and amplification (1000X) of the signal will be processed through a BioPac AcqKnowledge software system.

CONTACTS AND LOCATIONS:
Overall Officials: David G Behm, PhD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be available upon request to the individual. Anonymized data of the group will be available as supplementary material upon submission to a journal.